CLINICAL TRIAL: NCT07199517
Title: Catalyzing Cigarette Smoking Cessation Through Harm Reduction Sampling Among People Unmotivated to Quit
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: UPCC18025; 1R01CA302758-01 (NIH); 858599 (Other: University of Pennsylvania IRB)
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Cigarette Smoking; Tobacco Use; Cigarette Smoking Behavior
Keywords: cigarette smoking; harm reduction; sampling; nicotine replacement
MeSH Terms: conditions — Cigarette Smoking; Tobacco Use; Harm Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Harm Reduction Products (HRP) (Experimental): Participants randomized to HRP will try and rate ECIGS, IQOS, and ONPS during 3 virtual visits, and receive a 4-week supply of their preferred HRP (ECIGS, IQOS, or ONPs) for the sampling period.
  Interventions: Other: HRP Sampling period
- Nicotine Patch and Lozenge (NPL) (Active Comparator): Participants randomized to NPL will try a nicotine patch and nicotine lozenge during 1 virtual lab visit and will receive a 4-week supply of nicotine patches and lozenges for the sampling period.
  Interventions: Other: NPL Sampling period

INTERVENTIONS:
Other: HRP Sampling period — During a 28-day sampling period, participants randomized to HRP are instructed to try their selected HRP (ECIGS, IQOS, or ONPs) and will complete daily e-diaries of cigarette smoking behavior and product uptake.
  Arms: Harm Reduction Products (HRP)
Other: NPL Sampling period — During a 28-day sampling period, participants randomized to NPL are instructed to try nicotine patches and nicotine lozenges and will complete daily e-diaries of cigarette smoking behavior and product uptake.
  Arms: Nicotine Patch and Lozenge (NPL)

SUMMARY:
This study aims to investigate harm-reduction sampling in a choice format versus medicinal nicotine sampling on smoking behavior, identify mechanisms of sampling's effects, and explore moderators of these effects among a national sample of people unmotivated to quit smoking. Participants will be randomized 2:1 to choose one of three harm-reduction products (ECIG, IQOS, ONP) versus a medicinal nicotine control condition (nicotine patch + lozenge, NPL), receive a 4-week starter product regimen, and then be followed for 6 months to assess use behavior.

DETAILED DESCRIPTION:
Catalyzing smoking behavior change among people unready or unmotivated to quit smoking (PUQS) has the potential to disrupt decades of smoking and toxicant exposure, drastically reducing smoking-attributable morbidity and mortality. Unfortunately, current smoking cessation treatment approaches are typically designed for people who are seeking treatment and ready to quit smoking, which is the minority of people who smoke. Harm reduction product sampling, an extension of medication sampling, is a pragmatic and scalable approach to proactively engage people in transitioning away from combustible cigarette smoking. Sampling does not rely on sufficient motivation to initiate smoking behavior change. Rather, targeting behaviors consistent with quitting smoking (e.g., use of a starter regimen) can fuel motivation and smoking behavior change. In the only harm reduction sampling study to date, we found that a 4-week supply of e-cigarettes produced significant changes in smoking behavior compared to a no-provision control condition. E-cigarette uptake was robust compared to studies of medication sampling where no use or underuse of smoking cessation medication hindered sustained abstinence. These findings, coupled with our recent research, highlighted that any single harm-reduction product is only reinforcing to a fraction of users, but reinforcing value is one of the most important predictors of transitioning away from combustible cigarettes. As such, offering a choice among products is critical to provide appealing options for people with differing preferences and fully test the public health benefits of harm-reduction sampling among PUQS. Three potential alternatives to combusted cigarettes - e-cigarettes (ECIGS), heated tobacco products (IQOS), and oral nicotine pouches (ONPs) - each have the potential to reach more people who smoke than smoking cessation medication, resulting in a greater population reduction in harm from combustible tobacco. We propose the first investigation of harm-reduction sampling versus medicinal nicotine sampling on PUQS smoking behavior, mechanisms of sampling's effects, and potential moderators of these effects. A national sample of PUQS (n= 472, defined as not being ready to quit in the next 30 days) will be recruited and randomized 2:1 to choose one of three harm-reduction products (ECIG, IQOS, ONPs) versus a medicinal nicotine control condition (nicotine patch + lozenge, NPL). Product choice among those randomized to harm reduction will be informed by trying each product after biochemically confirmed overnight smoking abstinence, allowing each participant to try individual products before selecting their preferred option. Upon product selection (or assignment to NPL), participants will receive a 4-week starter product regimen. The primary outcome measure is a biochemically verified 7-day point prevalence smoking abstinence at the 6-month follow- up, with a 3-month follow-up as a secondary endpoint. Secondary outcomes include a 24-hour quit attempt and a 50% cigarette reduction per day. The findings have the potential to fill a critical clinical gap, advance evidence- based harm reduction approaches, and reduce smoking-attributable morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

1. Able to communicate fluently in English (i.e., speaking, writing, and reading)
2. Male and female smokers who are > 21 years of age and self-report smoking at least 5 cigarettes (menthol and/or non-menthol) per day for at least the last 6 months.
3. Have a carbon monoxide (CO) greater than or equal to 10 ppm
4. Not using any forms of nicotine regularly other than cigarettes.
5. Not interested in quitting smoking in the next 30 days.
6. Capable of giving written informed consent, including compliance with the requirements and restrictions listed in the combined consent and HIPAA form

Exclusion Criteria:

Smoking Behavior

1. Regular use of nicotine-containing products other than cigarettes (e.g., chewing tobacco, snuff, snus, cigars, e-cigs, IQOS, ONPS, etc.).
2. Current or impending (during the study period) enrollment or plans to enroll in a smoking cessation program.
3. Current use of smoking cessation medication.
4. Provide a CO breath test reading less than 10 ppm at Intake.

Alcohol and Drug

1. History of substance abuse (other than nicotine dependence) in the past 12 months.
2. Current alcohol consumption that exceeds 20 standard drinks/week.
3. Current use of recreational drugs (other than nicotine and cannabis)

Medical

1. Women, including all individuals assigned as "female" at birth, who are pregnant, breastfeeding, or planning a pregnancy over the duration of the study period.
2. Serious or unstable disease within the past year (e.g. cancer, uncontrolled hypertension, cardiovascular event).

Psychiatric

1. Lifetime history of schizophrenia or psychosis.

General Exclusion

1. Past, current, anticipated, or pending enrollment in another research program over the study period that could potentially impact subject safety, study data, and/or the study design as determined by the Principal Investigator.
2. Any medical condition, illness, disorder, adverse event (AE), or concomitant medication that could compromise participant safety or significantly impact study performance as determined by the Principal Investigator. Subjects may be deemed ineligible for any of the aforementioned reasons at any point throughout the study, as well as during the initial telephone screen.
3. Significant non-compliance with protocol and/or study design as determined by the Principal Investigator and/o. Subjects may be deemed ineligible at any point throughout the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 472 (Estimated)
Dates: Start 2026-01-12 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Smoking abstinence | 29 weeks
  Seven-day point prevalence smoking abstinence (CO < 5) will be measured at the 3-month (secondary endpoint) and 6-month follow-up (primary endpoint) via the valid and reliable TLFB procedure and biochemically verified through a CO < 5 ppm.

SECONDARY OUTCOMES:
Smoking reduction | 29 weeks
  Cigarette smoking rate and whether participants achieved a 50% change in cigarettes per day compared to their baseline smoking rate will be measured at the 3-month and 6-month follow-up via the valid and reliable TLFB procedure.
24-hour quit attempts | 29 weeks
  24-hour quit attempts and the number (count) of serious attempts to quit smoking, including those lasting greater than or equal to 24 hours, will be captured through diaries during the sampling period and the TLFB during follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Janet Audrain-McGovern, Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No